CLINICAL TRIAL: NCT02765438
Title: Lower Limb Muscle Activity During Task-specific Exercises With "BOBO"
Brief Title: Lower Limb Muscle Activity With "BOBO"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Isabella Shvartz, MD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOBO- HMO-CTIL
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BOBO (Experimental): Playing with the "BOBO" system.
  Interventions: Device: BOBO

INTERVENTIONS:
Device: BOBO — Each subject will play four games with the "BOBO" system.

SUMMARY:
Balance disorders are sometimes treated with exercises performed on unbalanced surfaces. The "BOBO" system allows connection of a standing platform attached to any of these surfaces, to a screen, where the user can control games with his or her body movements. In this study, the lower limb muscle activity of healthy individuals will be monitored during different games in order to assert the the ability of each game in strengthening certain muscle groups.

DETAILED DESCRIPTION:
Healthy subject will fill out a demographic questionnaire following the exercise they will fill out a subjective questionnaire for assessment of the exercise. Each subject will play 4 games using the "BOBO" while surface electrodes are placed on the gluteus max/medius, quadriceps, hamstring, peroneal ,tibialis anterior, gastrocnemius.

ELIGIBILITY:
Inclusion Criteria:

* Native Hebrew speaking

Exclusion Criteria:

* Familiar with the "BOBO" system
* Previous lower limb injuries
* Have a pacemaker
* Have neurological or vestibular deficiencies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Measuring the muscle activity using an Electromyography device | 2 hours
  The muscle activities of lower limb muscles using surface Electromyography device will be in units of volt.

IPD SHARING:
Plan to Share IPD: Undecided